CLINICAL TRIAL: NCT01985087
Title: A Phase I/ II Study of Hypofractionated Radiotherapy With Concurrent Temozolomide Followed by Adjuvant Temozolomide in Patients Over 70 Years Old With Newly Diagnosed Glioblastoma
Brief Title: A Study Using Radiation Therapy and Temozolomide to Treat Glioblastoma in Patients Over 70
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other)
Responsible Party: Principal Investigator, Adrianna H Masters, Assistant Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13.0538 BCC-NEU-13 GB70
Record Dates: First submitted 2013-10-10; First posted 2013-11-15 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiation Dose Hypofractionation; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hypofractionated radiotherapy and temozolomide (Experimental): All subjects will receive treatment as is a single arm study. Two weeks of combined hypofractionated radiotherapy with concurrent temozolomide followed by up to 6 cycles of adjuvant temozolomide treatment.
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: Temozolomide

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — Treatment of 3.4 Gy will be given daily 5 days per week over 2 weeks.
Drug: Temozolomide — During concomitant phase Temozolomide will be administered orally at 75 mg/m2 for 2 weeks concomitant with radiotherapy. During the adjuvant phase Temozolomide will be administered orally at 150 mg/m2 on days 1 through day 5 of each 28 day cycle for a maximum of 6 cycles.
  Other Names: Brand name Temodar

SUMMARY:
In this study we propose to determine outcomes of patients age 70 or older treated with radiation over 2 weeks given with temozolomide 75 mg/m2 daily during radiotherapy and as a post radiation treatment of 150 mg/m2 - 200 mg /m2 for 6 cycles or until the disease progresses.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically confirmed glioblastoma/gliosarcoma.
2. Tumor o6-methylguanine-DNA-methyltransferase promoter methylation status must be determined
3. Participants must not have had any prior therapy for glioblastoma multiforme including radiation or chemotherapy.
4. Participants must be > 70 years of age.
5. Participants must have life expectancy greater than 6 months.
6. Karnofsky performance status > 60 (ECOG < 2).
7. Patients must have normal organ and marrow function

   * Leukocytes > 3,000/microliter
   * Absolute neutrophil count > 1,500/microliter
   * Platelets > 100,000/microliter
   * Total bilirubin within normal institutional limits 12
   * aspartate aminotransferase test(SGOT)/alanine aminotransferase test(SGPT) < 2.5 X institutional upper limit of normal
   * Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Participants may not be receiving any other study agents.
2. Participants may not have had chemotherapy wafer placement at surgery.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide.
4. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
6. HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with temozolomide. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients who stop treatment due to Common Terminology Criteria for Adverse Events (CTCAE) grade 3 or above toxicities.. | baseline, 14-28 days post-surgery, 4 weeks post chemo-radiation therapy, 1, 2, 3, 4, 5, and 6 months post Radiation Therapy
  If < 4 out of 10 patients in the initial analysis stop treatment due to toxicity it can proceed to phase II.
Overall survival | From date of intervention until the date of first documented disease progression or death, the date of study discontinuation (e.g. toxicity, PI decision) or death from any cause, whichever is first, assessed up to 100 months.
  Survival status will be collected after completion of chemo-radiation at minimum every 3 months for up to 12 months, then every 6 months until date of death.

SECONDARY OUTCOMES:
Estimate progression-free survival (PFS) | From date of intervention until the date of first documented disease progression or death, the date of study discontinuation (e.g. toxicity, PI decision) or death from any cause, whichever is first, assessed up to 100 months.
  Survival/Documentation of progressive disease status will be collected every 3 months post chemo-radiation up to 12 months, then every 6 months until death, or from the date of disease progression, the date of study discontinuation (e.g. toxicity, PI decision), or from the date of the last dose of study drug (concomitant or adjuvant) if no disease progression.
Tolerability (feasibility) of hypo-fractionated radiaton therapy and Temozolomide | From date of intervention until the date of first documented disease progression or death, the date of study discontinuation (e.g. toxicity, PI decision) or death from any cause, whichever is first, assessed up to 100 months.
  Quality of life will be measured by Fact-BR assessment.

OTHER OUTCOMES:
Explore association of Overall Survival (OS) and Progression Free Survival (PFS) with 06-methylguanine-DNA methyltransferase gene (MGMT) methylation status | From date of intervention until the date of first documented disease progression or death, the date of study discontinuation (e.g. toxicity, PI decision) or death from any cause, whichever is first, assessed up to 100 months.
  Survival/Documentation of progressive disease status will be collected 4-weeks post chemo-radiation therapy then every 3 months up to 12 months, then every 6 months until death, from either the date of disease progression, the date of study discontinuation (e.g. toxicity, PI decision), or from the date of the last dose of study drug (concomitant or adjuvant) if no disease progression.
Explore changes in quality of life (QOL) | 14-28 days after surgery then within 4 weeks from end of chemotherapy-radiation then 1,4, and 6 months post initiation of adjuvant treatment
  To explore changes in QOL measured by Functional Assessment of Cancer Therapy (FACT-BR) and its predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Shiao Woo, MD, Principal Investigator — James Graham Brown Cancer Center
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States